CLINICAL TRIAL: NCT06161506
Title: A Phase II Trial of Surface Electrical Stimulation for Urinary Incontinence in Men Treated for Prostate Cancer
Brief Title: Surface Electrical Stimulation for Urinary Incontinence in Men Treated for Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001713; 001713-C
Record Dates: First submitted 2023-12-01; First posted 2023-12-08 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12-19

CONDITIONS: Urinary Urge Incontinence; Stress Urinary Incontinence; Prostatic Hyperplasia
Keywords: Elidah Device; Urinary Incontinence; Prostate Cancer
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Incontinence, Stress; Prostatic Hyperplasia; Urinary Incontinence; Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1/Elidah Device (Experimental): Elidah device application.
  Interventions: Device: Elidah Device

INTERVENTIONS:
Device: Elidah Device — The Elidah device is a modified version of the FDA approved ELITONE device cleared for use in the treatment of female stress urinary incontinence. For the current study, only minor modifications have been implemented with respect to the shape of the electrode component, providing a contour better suited to fit the male anatomy.

SUMMARY:
Background:

Men who are treated for prostate cancer often develop urinary leakage (incontinence). An experimental device that uses electrical impulses to stimulate pelvic floor muscles and surrounding tissues may help.

Objective:

To see if the Elidah device can reduce urinary incontinence after prostate treatment.

Eligibility:

Men aged 18 years and older who have had moderate urinary incontinence for at least 6 months after treatment for prostate cancer.

Design:

Participants will be in the study for about 9 weeks. They will be screened. They will have a physical exam with urine tests.

The Elidah device consists of a Controller and a GelPad. The Controller sets the strength of electrical impulses. The GelPad is placed against the skin under the pelvis.

Participants will be given an Elidah device and taught how to use it at home.

They will use the device once a day for 20 minutes at a time; they will do this 5 days a week for 6 weeks.

Participants will complete a daily log. They will record the strength of electrical impulses (0-35); the number of incontinence episodes; the type of incontinence episode; and the number of used pads.

Participants will do a pad weight test. For 3 days before and 3 days after using the Elidah device, they will collect all of their used pads for each 24-hour period into a sealed plastic bag. They will also collect a second set of bags that contain dry versions of each product used.

Participants will have clinic visits after using the device for 3 weeks and after finishing the 6 weeks of treatment.

Participants will complete 15-minute questionnaires.

DETAILED DESCRIPTION:
Background:

* Urinary incontinence is a common side effect of prostate cancer therapy that can negatively impact the quality of life.
* Standard treatment includes an initial course of pelvic floor muscle exercises followed by surgical therapy if urinary incontinence persists.
* Although pelvic floor muscle exercises can be successful in reducing urinary incontinence, compliance with exercises is poor.
* The Elitone (registered trademark) device was recently cleared by the Food and Drug Administration (FDA) for use in women with stress urinary incontinence. This device provides a surface electrical muscle stimulation device designed to contract the pelvic floor muscles and has been shown to reduce incontinence in women using the product.
* Recently, the electrode component (GelPad) of the device has been adapted for use in men by the manufacturing company, Elidah. The male version of the device is named the Elidah device.

Objective:

-To describe the efficacy of the Elidah device on male urinary incontinence

Eligibility:

* Participants must be male.
* Participants must have a history of urinary incontinence for at least 6 months after prostate cancer treatment.
* Participants must have at least one of the following types of urinary incontinence:

  * stress urinary incontinence, defined as involuntary loss of urine on effort or physical exertion (e.g., sporting activities), or on sneezing or coughing;
  * urge urinary incontinence, defined as a compelling need to urinate, due to pain or an unpleasant sensation, that is difficult to defer.

Design:

* This is a phase II trial testing the efficacy of the Elidah device in people treated for prostate cancer with stress and/or urge urinary incontinence.
* Prior to treatment, participants will undergo baseline assessments including 24-hour pad weight testing and questionnaires relating to incontinence and quality of life.
* Participants will self-administer the Elidah device treatment for 20 minutes per day, 5 days per week during a 6-week period in the at-home environment. Participants will maintain a Daily Log to record usage of the Elidah device, urinary leaks, and use of pads during each week of treatment.
* Following 6 weeks of therapy, participants will undergo re-evaluation of symptoms and urinary incontinence via questionnaires and testing with the 24-hour pad weight test.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must be male.
* Participants must have a history of urinary incontinence for at least 6 months after local prostate cancer treatment.
* Participants must have at least one of the following types of urinary incontinence:

  * stress urinary incontinence, defined as involuntary loss of urine on effort or physical exertion (e.g., sporting activities) or on sneezing or coughing
  * urge urinary incontinence, defined as a compelling need to urinate, due to pain or an unpleasant sensation, that is difficult to defer.
* Participants must have moderate urinary incontinence defined as use of 1-4 pads per day by self-report at screening.
* Participants must be able to read and write in English.
* Age >= 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status <= 2.
* Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Change of therapy for prostate cancer planned during the study intervention.
* History or symptoms of urinary retention (not an exclusion if this occurred before prostatectomy), extra-urethral incontinence, overflow incontinence.
* Active urinary tract infection (UTI) at screening or history of recurrent urinary tract infections (>= 4 UTIs within the 12 months prior to the study treatment initiation).
* History of complete denervation of the pelvic floor.
* Severe obesity (body mass index [BMI] >35).
* Pelvic pain/painful bladder syndrome.
* Metal implant in the abdominal or pelvic area.
* History of chronic cough with ongoing symptoms
* An implanted cardiac device, history of untreated cardiac arrhythmia, or history of other heart problems.
* History of epilepsy.
* History of underlying neurologic/neuromuscular disorder that could contribute to urinary incontinence.
* Change in medications prescribed for urinary incontinence within 2 weeks prior to the study treatment initiation.
* Uncontrolled intercurrent illness evaluated by medical history and physical examination or social situations that would limit compliance with study requirements.

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
To describe the efficacy of the Elidah device treatment on male urinary incontinence | Baseline and within 2 weeks after completing treatment
  Percent decrease in 24-hour pad weight after treatment with the Elidah device.

SECONDARY OUTCOMES:
To assess the safety of the Elidah device in men with urinary incontinence | 3 week visit and end of treatment visit
  Frequency of adverse events among treated participants and reporting the results, by maximum grade of event and type of toxicity noted.
To assess alternative measures of efficacy of Elidah device on male urinary incontinence and bother | Baseline and at end of treatment visit
  Evaluated by the number of pads and number of leaks before and after treatment. The mean of the percent reduction in the number of pads used per day following treatment will be computed along with 95% confidence intervals.
To assess participant-reported outcomes of Elidah device use for male urinary incontinence | Baseline and at end of treatment visit
  The proportion of participants for which the I-QoL score improves by 2.5 points or more following six weeks of Elidah device use will be estimated. 95% confidence intervals for this proportion will be constructed.
To assess treatment compliance with the Elidah device | 3 week visit and end of treatment visit
  A test of binomial proportions will be performed to assess whether the treatment noncompliance rate is above the unacceptability threshold.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah E Citrin, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001713-C.html